CLINICAL TRIAL: NCT03216915
Title: FINGORHYMS - Effects of Fingolimod on Heart Rhythm and Heart Rate Variability in Patients With Multiple Sclerosis
Brief Title: Effects of Fingolimod on Heart Rhythm and Heart Rate Variability in Patients With Multiple Sclerosis
Acronym: FINGORHYMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV5273
Record Dates: First submitted 2017-06-22; First posted 2017-07-13 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
Keywords: Heart Rhythm; Fingolimod; autonomic nervous system; Effects of Medicinal Substance
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Gilenya®; Novartis Pharmaceuticals Corporation — This is a prospective cohort-based study. Eligible are all patients planned for a treatment with fingolimod at the Hamburg University Hospital who are willing and able to participate in an observational study.
  Other Names: Fingolimod

SUMMARY:
The current study sought to prolong the observational interval after initiating medication with fingolimod and to measure the long-term effects of fingolimod on HR and HRV as an indicator of autonomic nervous system function in patients with RR-MS.

DETAILED DESCRIPTION:
Fingolimod (Gilenya®; Novartis Pharmaceuticals Corporation, East Hanover, NJ, USA) is a novel oral disease-modifying therapy that acts as a sphingosine-1-phosphate (S1P) receptor agonist and reduces the recirculation of lymphocytes to blood and peripheral tissues, including inflammatory lesions.

A critical part of fingolimod therapy still remains in the screening and initiation phases because of the risk of cardiac events. It is well known that the first dose of fingolimod is associated with a decrease in heart rate (HR) and slowing of atrioventricular (AV) conduction. Patients were continuously observed for a minimum of 6 hours after taking fingolimod. Because resurgence of heart rate began at 6 hours, the actual recommendation for observation is only 6 hours. Data about the effect of fingolimod after this time period is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent in accordance with Good Epidemiological Practice and local legislation
* Individuals over the age of 18 years
* Patients with relapsing-remitting forms of multiple sclerosis who were considered eligible for fingolimod treatment on a clinical basis.

Exclusion Criteria:

* Insufficient knowledge of the German language (not able to understand and write the German language)
* Physical or psychological incapability to take part in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing-remitting forms of multiple sclerosis who were considered eligible for fingolimod treatment on a clinical basis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of AF | 6 months follow up
  Recurrence of sustained atrial fibrillation (>30 seconds) after atrial fibrillation ablation

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, Principal Investigator — University Medical Hospital Hamburg-Eppendorf
Locations (1):
- University Medical Hospital Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided